CLINICAL TRIAL: NCT02421341
Title: Mechanisms of Altered Ventilatory Control in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas P. Olson, M.S., Ph.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-005318
Record Dates: First submitted 2015-02-25; First posted 2015-04-20 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
Keywords: Heart, Cardiovascular; Pulmonary; Skeletal Muscle; Exercise
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Fentanyl; Analgesics, Opioid; Catheters; Exercise; Respiratory Physiological Phenomena; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug - Fentanyl (Experimental): Study visit 1 you will be asked to get a blood draw, DEXA bone scan, perform pulmonary function tests, and exercise on a stationary bike at maximal exertion while breathing into a mouth piece. Study visits 2 and 3 you will be asked to again exercise at maximal exertion while breathing into a mouth piece. During these two visits you will be receiving an intrathecal injection of either fentanyl or placebo, randomly selected and you will be blinded as to which you are receiving. Catheters will also be placed in an artery in your arm and a vein in your leg, helping us to measure blood flow, blood pressure and draw blood. You will also perform a chemosensitivity test, breathing in and out your own air, after you are done exercising.
  Interventions: Drug: Fentanyl; Procedure: Catheters; Other: Exercise; Radiation: DEXA; Other: Pulmonary Function Tests; Other: Blood Draw; Other: Chemosensitivity Test
- Placebo (Placebo Comparator): Study visit 1 you will be asked to get a blood draw, DEXA bone scan, perform pulmonary function tests, and exercise on a stationary bike at maximal exertion while breathing into a mouth piece. Study visits 2 and 3 you will be asked to again exercise at maximal exertion while breathing into a mouth piece. During these two visits you will be receiving an intrathecal injection of either fentanyl or placebo, randomly selected and you will be blinded as to which you are receiving. Catheters will also be placed in an artery in your arm and a vein in your leg, helping us to measure blood flow, blood pressure and draw blood. You will also perform a chemosensitivity test, breathing in and out your own air, after you are done exercising.
  Interventions: Procedure: Catheters; Other: Exercise; Radiation: DEXA; Other: Pulmonary Function Tests; Other: Blood Draw; Other: Chemosensitivity Test; Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl — During study visits 2 and 3 you will receive an intrathecal (fluid filled space surrounding the spinal cord) injection of either fentanyl or placebo (saline). Fentanyl is an opiate (narcotic) drug and a common medication, however the way fentanyl is being used in this study is considered investigational.
  Other Names: Analgesic, Opioid
  Arms: Drug - Fentanyl
Procedure: Catheters — A catheter (small plastic tube placed in a blood vessel) will be placed in an artery in your arm and a second catheter will be placed in a vein in your leg. Local anesthetic will be used to minimize discomfort. These catheters will allow us to measure blood pressure, leg blood flow and draw blood.
Other: Exercise — You will be asked to exercise, ride a stationary bike, at maximal exertion.
Radiation: DEXA — During study visit one you will have a DEXA scan. This procedure requires you to lie on a table while a small x-ray tube passes under your body.
Other: Pulmonary Function Tests — During study visit one you will be asked to perform 5 different breathing tests to help us better understand your lung function.
Other: Blood Draw — You will have approximately 350 mls (1.25 cups) of blood drawn during the duration of this study.
Other: Chemosensitivity Test — Using a bag you breath in and out your own air.
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is being done because the investigators are trying to understand how feedback from the muscles can influence your blood pressure and breathing during exercise, and if the investigators can reduce this response in heart failure patients. The investigators are also trying to determine ways to improve tolerance to exercise in heart failure patients.

DETAILED DESCRIPTION:
If you are enrolled in this study the investigators will ask you to make 3 separate study visits.

During study visit 1 you will be asked to get a blood draw, DEXA bone scan, perform pulmonary function tests, and exercise on a stationary bike at maximal exertion while breathing into a mouth piece.

During study visits 2 and 3 you will be asked to again exercise at maximal exertion while breathing into a mouth piece. However, during these two visits you will be receiving an intrathecal injection of fentanyl one day and placebo the other day, randomly selected and you will be blinded as to which you are receiving. A catheter will also be placed in an artery in your arm and a vein in your leg, which will help us to measure blood flow, blood pressure and draw blood when need be. The investigators will also ask you to perform a brief chemosensitivity test, breathing in and out your own air, after you are done exercising.

ELIGIBILITY:
Inclusion Criteria (Heart Failure Patients):

* History of ischemic or idiopathic dilated cardiomyopathy
* New York Heart Association class 1-3
* No history of dangerous arrhythmia's
* Not pacemaker dependent
* Body Mass Index less than or equal to 35 kg/m
* Current non-smokers with less than 15 pack year history
* Non-pregnant women
* Individuals who are able to exercise without orthopedic limitations
* All patients will be managed by their primary care physician or cardiologist prior to enrollment to ensure inclusion and exclusion criteria have been satisfied and participation in exercise testing is safe.

Control Participants:

* Will be matched for age, gender, height and weight and will have no history of cardiovascular related abnormalities.
* Body Mass Index less than 35 kg/m
* Current non-smokers with less than 15 pack year history
* Non-pregnant women
* Individuals who are able to exercise without orthopedic limitations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-07; Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Capacity to exercise (gas exchange analysis, borg scale questions, and medical doctor supervision) | An expected average of 4 hours.
  Participants will be monitored during the duration of their exercise by gas exchange analysis, borg scale questions, and medical doctor supervision.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Olson, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - Saint Marys Hospital, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials